CLINICAL TRIAL: NCT01036685
Title: Cognitive Task Development and Implementation for Functional MRI Studies
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903379; 03-DA-N379
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-05

CONDITIONS: Drug Abuse; Nicotine Dependence
Keywords: Task Development; Natural History; fMRI; Cognition; Affect
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- 379-bench-control: healthy control who will only do behavioral tasks
- 379-bench-other-psych-diagnosis: someone with a DSM-V disorder, stable and in treatment (i.e., no medication changes in the previous four weeks and a clearly identified treating psychiatrist) who will only do behavioral tasks
- 379-bench-smoker: daily smoker of tobacco cigarettes for at least one year (excluding quit attempts) who will only do behavioral tasks
- 379-bench-user: someone with a DSM-V substance use disorder on a substance other than nicotine who will only do behavioral tasks
- 379-control: healthy control who can do MRI
- 379-other-psych -diagnosis: someone with a DSM-V disorder, stable and in treatment (i.e., no medication changes in the previous four weeks and a clearly identified treating psychiatrist) who can do MRI
- 379-smoker: daily smoker of tobacco cigarettes for at least one year (excluding quit attempts) who can do MRI
- 379-user: someone with a DSM-V substance use disorder on a substance other than nicotine who can do MRI

SUMMARY:
Background:

* Drugs of abuse have effects on mood, behavior, thinking, and decision making that may encourage people to continue using them and make it difficult for them to stop. Researchers who study these effects are interested in developing new tests to evaluate how drugs and drug use affect different areas of the brain.
* Magnetic resonance imaging (MRI) scans allow researchers to study brain activity and changes to brain function. When specific psychological tests are performed during functional MRI (fMRI) scans, researchers can examine the effects of drug use on the brain. By developing and testing new procedures for fMRI studies, more information can be obtained on brain function and activity in drug-using and non-drug-using individuals, and this information can help develop new treatments and therapies for substance abuse.

Objectives:

- To develop, assess and refine of cognitive and affective tasks and determination of their practical feasibility and efficacy for both MRI and non-MRI application.

Eligibility:

* Healthy volunteers between 18 and 65 years of age who are willing to undergo MRI scanning.
* Both drug-using and non-drug-using individuals will be selected for this study.

Design:

* Before the start of the study, participants may complete as assessment of medical and psychological history, and provide information about past or current drug use. Researchers will introduce the tasks to be performed and may have participants practice the tasks.
* During the study, participants will be asked to do one or more tasks selected by the researchers. The tasks may be performed on a computer in an MRI machine, and may involve receiving rewards (such as money or sips of juice) for actions, memory and reaction-time tests, or other tests that involve responding to instructions on the screen.
* Participants will receive compensation for their participation in the study, including hourly compensation for individual visits.

DETAILED DESCRIPTION:
Objective: Drugs of abuse have cognitive and affective effects that may contribute to the inception and maintenance of their use. In order to measure these effects, psychological tests suitable for use both in and outside the fMRI scanner need to be developed and validated. Thus, the objective of this protocol is to allow for the development, assessment and refinement of cognitive and affective tasks and determination of their practical feasibility and efficacy for both MRI and non-MRI application.

Study Population: This minimal-risk protocol will employ volunteer participants aged 18-65, who must be generally healthy. In order to ensure applicability to relevant groups, both drug and nondrug using volunteers as well as those recruited from clinical populations will be used to validate task design and parameters.

Design: Participants may pilot tasks outside and/or inside the MRI scanner, depending on the aspects of task development requiring verification. Tasks developed de novo will undergo both steps. Modifications to previously published MRI tasks may require only one of the steps. Upon their successful verification, specific experimental manipulations will be performed under separate, hypothesis driven protocols.

Outcome measures: Our goal is to determine if the tasks developed reliably and appropriately measure specific cognitive constructs and behaviors thought to be associated with specific brain systems, if they yield measurable and interpretable fMRI results.

ELIGIBILITY:
* INCLUSION CRITERIA:

Bench Only Phase (no MRI)

Participants will be considered for one of three categories: 379-bench-control, 379-bench-smoker/vaper, 379-bench-user. Vapers will be admitted to experiments involving smoking cues (with cues specific to vaping) because it has been shown that responses to vaping cues are very similar to responses to smoking cues and can be lumped together in analyses.

Participant must meet the following inclusion criteria for the Bench Only Phase:

1. Between the ages of 18-65.
2. All subjects must be able to provide informed consent/assent.
3. Additional criteria for specific populations:

   1. 379-bench-smoker/vaper: regular smoker of tobacco cigarettes or nicotine vaper with a urine cotinine level corresponding to nicotine user status for the specific test being used (typically corresponding to a urine cotinine above about 200 ng/ml) and have been smoking or vaping consistently for at least one year (excluding quit attempts)
   2. 379-bench-user: DSM-V substance use disorder on a substance other than nicotine.

EXCLUSION CRITERIA:

Bench Only Phase (Does not require MRI. Task requires gathering of accurate behavioral data).

1. History of neurologic injury including but not limited to CVA, CNS tumor, or head trauma with persistent sequelae. Assessment tool: pre-screen survey and medical history.

   Rationale: Neurologic injury is likely to impair performance on the range of tasks to be piloted under this protocol.
2. Current use of psychoactive medications likely to affect the performance of the task under consideration, unless required for the psychiatric disorder for which participants in the 379-user and 379-other-psych-diagnosis subcategories are being treated. Assessment tool: pre-screen survey, medical history. Rationale: certain psychoactive medications may alter performance on the range of tasks to be piloted under this protocol.
3. Cognitive impairment. Assessment tool: self report of extended placement in special education classes for learning problems, history of specific learning disability or mental retardation. Rationale: Cognitive impairment is likely to impair performance on the range of tasks to be piloted under this protocol and may impair ability to tolerate the procedures.
4. Current major mood, anxiety or psychotic disorder with symptoms severe enough to impair ability to participate (unless task is being evaluated in a specific clinical population). Assessment tool: self report, medical history. Rationale: Current major mood or psychotic disorders with poorly controlled symptoms may impair performance on the range of tasks to be piloted under this protocol and may impair ability to tolerate the procedures.
5. Non-English speaking. Assessment tool(s): self-report. Rationale: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing study procedures. The inability to effectively communicate safety procedures in a language other than English could compromise the safety of non-English speaking participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects must be between the ages of 18-65 and be generally healthy. (Please note that references to adults in this protocol refers to those age 18 and older). Depending on the task being developed and specific task goals, they may have a substance use disorder or have no history of substance use.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2005-05-22 (Actual)

PRIMARY OUTCOMES:
To determine if the tasks reliably and appropriately measure specific cognitive constructs and behaviors thought to be associated with specific brain systems and, also if they yield measurable and interpretable fMRI results. | each visit
  1. To derive the parameters necessary to determine the reliability and validity of cognitive tasks.2. To determine the ability of various control and target populations to perform the tasks appropriately in and out of the MRI scanner.3. To determine the task parameters optimal for the activation of specific brain regions when employed during fMRI scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Ross, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share raw data from the study as this is a task development protocol in which the objective is the development, assessment and refinement of cognitive and affective tasks and determination of their practical feasibility and efficacy for both MRI and non-MRI application for future protocols.